CLINICAL TRIAL: NCT03256786
Title: Effects of Preanesthetic Forced Air Warming and Administration of Warmed Intravascular Fluid on Preventing Hypothermia and Shivering During Cesarean Delivery Under Spinal Anesthesia
Brief Title: Effects of Preanesthetic Forced Air Warming and Administration of Warmed Intravascular Fluid
Status: Completed | Type: Observational
Sponsor: Hallym University Kangnam Sacred Heart Hospital (Other)
Responsible Party: Principal Investigator, Choi Eun MI, Clinical Professor, Hallym University Kangnam Sacred Heart Hospital
Other Study IDs: kangnamAN
Record Dates: First submitted 2017-08-15; First posted 2017-08-22 (Actual); Last update posted 2019-02-27 (Actual); Status verified 2019-02

CONDITIONS: Pregnancy
Keywords: cesarean delivery with spinal anesthesia; Hypothermia and shivering; Active warming
MeSH Terms: conditions — Hypothermia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Active warming: preoperative 15 min of surface warming using a forced air warmer before spinal anesthesia and coloading of warmed intravenous fluid
  Interventions: Behavioral: Prewarming using forced air warmer, warmed intravenous fluid
- Control: no preoperative warming and room temperature intravenous fluid

INTERVENTIONS:
Behavioral: Prewarming using forced air warmer, warmed intravenous fluid — Combined modality active warming consisting of preoperative 15 min of surface warming using a forced air warmer before spinal anesthesia and coloading of warmed intravenous fluid in active warming group
  Groups: Active warming

SUMMARY:
The majority of women (> 60%) developed hypothermia and shivering during cesarean delivery. Core hypothermia may be associated with a number of adverse outcomes in patients, including shivering, wound infection, coagulopathy, increased blood loss and transfusion requirements, decreased metabolism and prolonged recovery. Shivering can result in interference with monitoring, increased tension on wound edges, and increased oxygen consumption.

A previous study has shown several modalities to prevent hypothermia and shivering in patients undergoing cesarean delivery with spinal anesthesia. But, single modality intervention have shown marginal or no efficacy.

Neuraxial anesthesia reduces the threshold for vasoconstriction and shivering. It often also produces a lower body sympathectomy that provokes a core to peripheral redistribution of body heat. It is difficult to treat the core to peripheral redistribution of body heat. However redistribution can be prevented by preanesthetic cutaneous warming. Prewarming hardly changes core temperature that remains well regulated, but it markedly increases peripheral tissue heat content. As a result, prewarming reduces the core to peripheral tissue temperature gradient and the propensity for redistribution after the induction of anesthesia.

We therefore hypothesized that Combined modality active warming consisting of preoperative 15 min of surface warming using a forced air warmer before spinal anesthesia and coloading of warmed intravenous fluid might reduce perioperative hypothermia and shivering in women undergoing cesarean delivery. Additionally, We tested the hypothesis that maintaining maternal normothermia increases newborn temperature and Apgar scores.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for cesarean delivery under spinal anesthesia
* The American Society of Anesthesiologists physical status class one or two
* female between 20 and 45

Exclusion Criteria:

* Patients with heart disease
* Patients with infectious disease
* Patients with coagulopathy
* Patients with a drug allergy
* In case of switching to general anesthesia
* Patients BMI under 18.5 or over 31

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients scheduled for cesarean delivery under spinal anesthesia
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2017-07-12 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2018-04-30 (Actual)

PRIMARY OUTCOMES:
incidence of hypothermia and shivering | immediately after arrival at the postanesthesia care unit

SECONDARY OUTCOMES:
temperature of newborn | immediately after delivery of newborn

CONTACTS AND LOCATIONS:
Overall Officials: Eun Mi Choi, MD, Study Director — Hallym University Kangnam Sacred Heart Hospital
Locations (1):
- Kangnam sacred heart hospital, Seoul, Yeongdeungpo-gu, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Carpenter L, Baysinger CL. Maintaining perioperative normothermia in the patient undergoing cesarean delivery. Obstet Gynecol Surv. 2012 Jul;67(7):436-46. doi: 10.1097/OGX.0b013e3182605ccd. PMID 22926250
- [Result] Kurz A, Sessler DI, Lenhardt R. Perioperative normothermia to reduce the incidence of surgical-wound infection and shorten hospitalization. Study of Wound Infection and Temperature Group. N Engl J Med. 1996 May 9;334(19):1209-15. doi: 10.1056/NEJM199605093341901. PMID 8606715
- [Result] Frank SM, Fleisher LA, Breslow MJ, Higgins MS, Olson KF, Kelly S, Beattie C. Perioperative maintenance of normothermia reduces the incidence of morbid cardiac events. A randomized clinical trial. JAMA. 1997 Apr 9;277(14):1127-34. PMID 9087467
- [Result] Schmied H, Kurz A, Sessler DI, Kozek S, Reiter A. Mild hypothermia increases blood loss and transfusion requirements during total hip arthroplasty. Lancet. 1996 Feb 3;347(8997):289-92. doi: 10.1016/s0140-6736(96)90466-3. PMID 8569362
- [Result] Knobel RB, Wimmer JE Jr, Holbert D. Heat loss prevention for preterm infants in the delivery room. J Perinatol. 2005 May;25(5):304-8. doi: 10.1038/sj.jp.7211289. PMID 15861196
- [Result] Watkinson M. Temperature control of premature infants in the delivery room. Clin Perinatol. 2006 Mar;33(1):43-53, vi. doi: 10.1016/j.clp.2005.11.018. PMID 16533632
- [Result] Butwick AJ, Lipman SS, Carvalho B. Intraoperative forced air-warming during cesarean delivery under spinal anesthesia does not prevent maternal hypothermia. Anesth Analg. 2007 Nov;105(5):1413-9, table of contents. doi: 10.1213/01.ane.0000286167.96410.27. PMID 17959975
- [Result] Yokoyama K, Suzuki M, Shimada Y, Matsushima T, Bito H, Sakamoto A. Effect of administration of pre-warmed intravenous fluids on the frequency of hypothermia following spinal anesthesia for Cesarean delivery. J Clin Anesth. 2009 Jun;21(4):242-8. doi: 10.1016/j.jclinane.2008.12.010. Epub 2009 Jun 6. PMID 19502035
- [Result] Cobb B, Cho Y, Hilton G, Ting V, Carvalho B. Active Warming Utilizing Combined IV Fluid and Forced-Air Warming Decreases Hypothermia and Improves Maternal Comfort During Cesarean Delivery: A Randomized Control Trial. Anesth Analg. 2016 May;122(5):1490-7. doi: 10.1213/ANE.0000000000001181. PMID 26895002
- [Result] Horn EP, Schroeder F, Gottschalk A, Sessler DI, Hiltmeyer N, Standl T, Schulte am Esch J. Active warming during cesarean delivery. Anesth Analg. 2002 Feb;94(2):409-14, table of contents. doi: 10.1097/00000539-200202000-00034. PMID 11812709
- [Result] Matsukawa T, Sessler DI, Christensen R, Ozaki M, Schroeder M. Heat flow and distribution during epidural anesthesia. Anesthesiology. 1995 Nov;83(5):961-7. doi: 10.1097/00000542-199511000-00008. PMID 7486181
- [Result] Matsukawa T, Sessler DI, Sessler AM, Schroeder M, Ozaki M, Kurz A, Cheng C. Heat flow and distribution during induction of general anesthesia. Anesthesiology. 1995 Mar;82(3):662-73. doi: 10.1097/00000542-199503000-00008. PMID 7879935
- [Result] Rajek A, Greif R, Sessler DI. Effects of epidural anesthesia on thermal sensation. Reg Anesth Pain Med. 2001 Nov-Dec;26(6):527-31. doi: 10.1053/rapm.2001.25924. PMID 11707791
- [Result] Chung SH, Lee BS, Yang HJ, Kweon KS, Kim HH, Song J, Shin DW. Effect of preoperative warming during cesarean section under spinal anesthesia. Korean J Anesthesiol. 2012 May;62(5):454-60. doi: 10.4097/kjae.2012.62.5.454. Epub 2012 May 24. PMID 22679543
- [Derived] Jun JH, Chung MH, Jun IJ, Kim Y, Kim H, Kim JH, Choi YR, Choi EM. Efficacy of forced-air warming and warmed intravenous fluid for prevention of hypothermia and shivering during caesarean delivery under spinal anaesthesia: A randomised controlled trial. Eur J Anaesthesiol. 2019 Jun;36(6):442-448. doi: 10.1097/EJA.0000000000000990. PMID 30985539